CLINICAL TRIAL: NCT00320216
Title: A Phase II, Randomized, Double-blind, Placebo-controlled, Parallel Study of Single and Multiple Dose Regimens With Subcutaneous CNTO 1275 (Human Monoclonal Antibody to IL-12) in Subjects With Moderate to Severe Psoriasis
Brief Title: A Safety and Effectiveness Study of CNTO 1275 in Patients With Moderate to Severe Plaque-type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005416; C0379T04 (Other: Centocor); NCT00322998 (obsolete NCT alias)
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Results first posted 2012-12-19 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-03

CONDITIONS: Psoriasis
Keywords: Psoriasis; CNTO 1275; Ustekinumab; Stelara; Interleukin-12; IL-12; Interleukin-23; IL-23
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group I (Placebo) (Placebo Comparator): Patients in the placebo group will receive placebo at Weeks 0, 1, 2, 3, and 16. At week 20, all patients will receive a single dose of ustekinumab 90 mg.
  Interventions: Drug: Placebo
- Group II (Ustekinumab 45 mg) (Experimental): Patients will receive single dose ustekinumab at Week 0 and placebo at Weeks 1, 2, and 3. At Week 16, patients with Physician's Global Assessment (PGA) greater than or equal to 3 will receive ustekinumab 45 mg. At week 20, all patients will receive placebo.
  Interventions: Drug: Ustekinumab; Drug: Placebo
- Group III (Ustekinumab 90 mg) (Experimental): Patients will receive 90 mg single dose ustekinumab at Week 0 and placebo at Weeks 1, 2, and 3. At Week 16 patients with PGA greater than or equal to 3 will receive ustekinumab 90 mg. At week 20, all patients will receive placebo.
  Interventions: Drug: Ustekinumab; Drug: Placebo
- Group IV (Experimental): Patients will receive 45 mg of ustekinumab at Weeks 0, 1, 2, and 3. At Week 16, patients with Physician's Global Assessment (PGA) greater than or equal to 3 will receive ustekinumab 45 mg. At week 20, all patients will receive placebo.
  Interventions: Drug: Ustekinumab
- Group V (Experimental): Patients will receive 90 mg of ustekinumab at Weeks 0, 1, 2, and 3. At Week 16 patients with Physician's Global Assessment (PGA) greater than or equal to 3 will receive ustekinumab 90 mg. At week 20, all patients will receive placebo.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Patients will receive subcutaneous injections of ustekinumab (45 or 90 mg).
  Other Names: CNTO 1275
  Arms: Group II (Ustekinumab 45 mg); Group III (Ustekinumab 90 mg); Group IV; Group V
Drug: Placebo — Patients in the placebo group will receive placebo medication.
  Arms: Group I (Placebo); Group II (Ustekinumab 45 mg); Group III (Ustekinumab 90 mg)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of initial single and multiple subcutaneous injections of CNTO 1275 in the treatment of patients with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), double blind (neither physician nor patient knows the treatment that the patient receives), parallel-group, multicenter study to determine the effectiveness and safety of two different doses of CNTO 1275 administered subcutaneously one time or as multiple doses as compared with placebo in patients with moderate to severe plaque-type psoriasis (the most common type of psoriasis). The dose of CNTO 1275 will be 45 or 90 mg administered subcutaneously once or as four weekly doses. Patients who inadequately respond to their treatment may receive one additional dose. Patients will be monitored for the safety throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have had a diagnosis of plaque-type psoriasis at least 6 months
* Plaque-type psoriasis covering at least 10% of total body surface areas
* Psoriasis area-and-severity index score of 12 or greater
* Considered by treating dermatologist to be a candidate for phototherapy or systemic treatment of psoriasis
* Women of childbearing potential and all men must agree to use adequate birth control measures
* Have no history of latent or active tuberculosis

Exclusion Criteria:

* Currently have nonplaque forms of psoriasis or drug-induced psoriasis
* Women who are pregnant or nursing, or men and women planning pregnancy while enrolled in the study
* Patients who have a history of chronic or recurrent infectious disease or who have or have had a serious infection requiring hospitalization or intravenous antibiotics within the previous 2 months
* Patients who have or ever have had a nontuberculous mycobacterial infection or opportunistic infection
* Patients known to be infected with human immunodeficiency virus, hepatitis B, or hepatitis C
* Patients who have current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease
* Have any known malignancy or have a history of malignancy within the previous 5 years (with the exception of basal cell carcinoma of the skin that has been treated with no evidence of recurrence)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2003-11; Primary Completion 2004-06 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Derived] Ghosh S, Gensler LS, Yang Z, Gasink C, Chakravarty SD, Farahi K, Ramachandran P, Ott E, Strober BE. Ustekinumab Safety in Psoriasis, Psoriatic Arthritis, and Crohn's Disease: An Integrated Analysis of Phase II/III Clinical Development Programs. Drug Saf. 2019 Jun;42(6):751-768. doi: 10.1007/s40264-019-00797-3. PMID 30739254
- [Derived] Krueger GG, Langley RG, Leonardi C, Yeilding N, Guzzo C, Wang Y, Dooley LT, Lebwohl M; CNTO 1275 Psoriasis Study Group. A human interleukin-12/23 monoclonal antibody for the treatment of psoriasis. N Engl J Med. 2007 Feb 8;356(6):580-92. doi: 10.1056/NEJMoa062382. PMID 17287478

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 320 participants from 45 sites in North America were randomized to receive either Ustekinumab or placebo.
Groups:
- Placebo (CP): Controlled period (Week 0-20) - receiving placebo at Weeks 0, 1, 2, 3 and 16.
- Ustekinumab 45 mg (CP): Controlled period (Week 0-20) - receiving ustekinumab 45 mg at Weeks 0. At week 16, participants with PGA >= 3 received ustekinumab 45 mg.
- Ustekinumab 90 mg (CP): Controlled period (Week 0-20) - receiving ustekinumab 90 mg at Weeks 0. At week 16, participants with PGA >= 3 received ustekinumab 90 mg.
- Ustekinumab 45 mg Weekly for 4 Weeks (CP): Controlled period (Week 0-20) - receiving ustekinumab 45 mg at Weeks 0, 1, 2 and 3. At week 16, participants with PGA >= 3 received ustekinumab 45 mg.
- Ustekinumab 90 mg Weekly for 4 Weeks (CP): Controlled period (Week 0-20) - receiving ustekinumab 90 mg at Weeks 0, 1, 2 and 3. At week 16, participants with PGA >= 3 received ustekinumab 90 mg.
Period: Overall Study
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP) | Ustekinumab 45 mg Weekly for 4 Weeks (CP) | Ustekinumab 90 mg Weekly for 4 Weeks (CP)
Started | 64 | 64 (1 patient randomized but not treated was included as discontinued due to Other reason.) | 64 (1 patient randomized but not treated was included as discontinued due to Other reason.) | 64 | 64
Completed | 48 | 54 | 58 | 61 | 58
Not Completed | 16 | 10 | 6 | 3 | 6
Not completed — Adverse Event | 0 | 6 | 0 | 2 | 2
Not completed — Lack of Efficacy | 6 | 2 | 1 | 0 | 1
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0 | 0
Not completed — Other | 7 | 2 | 5 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Group I: Placebo: Participants received placebo at Weeks 0, 1, 2 and 3. At week 16, all participants received placebo regardless of Physician's Global Assessment (PGA). At week 20, all participants received a single dose of ustekinumab 90 mg.
- Group II: Ustekinumab 45 mg: Participants received ustekinumab 45 mg at Week 0 followed by placebo at Weeks 1, 2 and 3. At week 16, participants who had a Physician's Global Assessment (PGA) >=3 received 45 mg ustekinumab and participants with a PGA<3 received placebo. At week 20, all participants received placebo.
- Group III: Ustekinumab 90 mg: Participants received ustekinumab 90 mg at Week 0 followed by placebo at Weeks 1, 2 and 3. At week 16, participants who had a Physician's Global Assessment (PGA) >=3 received 90 mg ustekinumab and participants with a PGA<3 received placebo. At week 20, all participants received placebo.
- Group IV: Ustekinumab 45 mg Weekly for 4 Weeks: Participants received ustekinumab 45 mg at Weeks 0, 1, 2 and 3. At week 16, participants who had a Physician's Global Assessment (PGA) >=3 received 45 mg ustekinumab and participants with a PGA<3 received placebo. At week 20, all participants received placebo.
- Group V: Ustekinumab 90 mg Weekly for 4 Weeks: Participants received ustekinumab 90 mg at Weeks 0, 1, 2 and 3. At week 16, participants who had a Physician's Global Assessment (PGA) >=3 received 90 mg ustekinumab and participants with a PGA<3 received placebo. At week 20, all participants received placebo.
- Total: Total of all reporting groups
Arm/Group | Group I: Placebo | Group II: Ustekinumab 45 mg | Group III: Ustekinumab 90 mg | Group IV: Ustekinumab 45 mg Weekly for 4 Weeks | Group V: Ustekinumab 90 mg Weekly for 4 Weeks | Total
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 64 | 320
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Years | 44.0 (13.7) | 46.4 (14.2) | 45.5 (12.7) | 44.5 (12.2) | 44.3 (13.3) | 44.9 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 26 | 17 | 25 | 52 | 138
  Male | 46 | 38 | 47 | 39 | 12 | 182

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Psoriasis Area and Severity Index (PASI) 75% Improvement at Week 12
Description: Psoriasis Area and Severity Index (PASI)(0 [ best] -72 [worst]) score at Week 12. This is a test of how bad a person's psoriasis is. The combination of redness, scaling, and thickness, as well as overall body involvement determine the PASI score.
Time Frame: Week 12
Population: Intent to treat. All participants randomized were included in the analysis according to the assigned treatment groups. Participant is considered a non- responder if the participant has used any pre-specified prohibited medications or discontinued due to lack of efficacy.
Measure: Number; unit: Participants
Arm/Group | Group I: Placebo | Group II: Ustekinumab 45 mg | Group III: Ustekinumab 90 mg | Group IV: Ustekinumab 45 mg Weekly for 4 Weeks | Group V: Ustekinumab 90 mg Weekly for 4 Weeks
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 64
Participants | 1 | 33 | 38 | 43 | 52
Statistical Analysis 1: Comparison: Group I: Placebo vs Group V: Ustekinumab 90 mg Weekly for 4 Weeks; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi square test; Stratified by baseline weight [<=90kg vs > 90 kg]
Statistical Analysis 2: Comparison: Group I: Placebo vs Group IV: Ustekinumab 45 mg Weekly for 4 Weeks; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square; Stratified by baseline weight [≤ 90kg vs > 90 kg)]
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square; Stratified by baseline weight [≤ 90kg vs > 90 kg)]
Statistical Analysis 4: Comparison: Group I: Placebo vs Group II: Ustekinumab 45 mg; Null Hypothesis:No difference between any ustekinumab group and placebo at an overall significant level of 0.05. Sample Size: With 300 participants (60 in each treatment group), simulation studies were conducted to calculate the power to detect a treatment difference in primary endpoint between ustekinumab groups and placebo using a CMH test with stratification by baseline weight [≤ 90kg vs > 90 kg). For all the scenarios evaluated, the power is >99% at an overall significance level of 0.05; Test type: Superiority or Other; p < 0.01, Cochran-Mantel-Haenszel (CMH) chi square — To control for the multiplicity for the primary endpoint analysis, the 4 pairwise comparisons between ustekinumab groups and placebo were performed sequentially at alpha = 0.05. The order of testing was prespecified from high to low doses; Stratified by baseline weight [≤ 90kg vs > 90 kg)]

2. Secondary Outcome: Number of Participants Who Achieved Physician's Global Assessment (PGA) Score of Clear (1) or Excellent (2) at Week 12
Description: Number of participants achieving a physician global assessment (PGA)(1 [best] to 6 [worst]) score of clear or excellent at Week 12. The PGA is used to determine the participants psoriasis lesions overall at a given time point. Overall lesions will be graded for induration, erythema, and scaling. The sum of the 3 scales will be divided by 3 to obtain a final PGA score.
Time Frame: Week 12
Population: Participants were included in the analysis according to the assigned treatment groups. Participant is considered a non- responder if the participant has used any pre-specified prohibited medications or discontinued due to lack of efficacy. Other missing data were not imputed.
Measure: Number; unit: Participants
Arm/Group | Group I: Placebo | Group II: Ustekinumab 45 mg | Group III: Ustekinumab 90 mg | Group IV: Ustekinumab 45 mg Weekly for 4 Weeks | Group V: Ustekinumab 90 mg Weekly for 4 Weeks
Number analyzed (Participants) | 64 | 63 | 64 | 64 | 64
Participants | 0 | 32 | 34 | 46 | 53
Statistical Analysis 1: Comparison: Group I: Placebo vs Group V: Ustekinumab 90 mg Weekly for 4 Weeks; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square; Stratified by baseline weight [≤ 90kg vs > 90 kg)]
Statistical Analysis 2: Comparison: Group I: Placebo vs Group IV: Ustekinumab 45 mg Weekly for 4 Weeks; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square; Stratified by baseline weight [≤ 90kg vs > 90 kg)]
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square
Statistical Analysis 4: Comparison: Group I: Placebo vs Group II: Ustekinumab 45 mg; Null Hypothesis: No difference between any ustekinumab group and placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square; Stratified by baseline weight [≤ 90kg vs > 90 kg)]

3. Secondary Outcome: Number of Participants Who Achieved Psoriasis Area Severity Index (PASI) 75% Improvement at Week 32
Description: Psoriasis Area and Severity Index (PASI)(0 [ best] -72 [worst]) score at Week 32 for participants who were not retreated at Week 16. This is a test of how bad a person's psoriasis is. The combination of redness, scaling, and thickness, as well as overall body involvement determine the PASI score.
Time Frame: Week 32
Population: as for outcome 2
Measure: Number; unit: Particpants
Arm/Group | Group I: Placebo | Group II: Ustekinumab 45 mg | Group III: Ustekinumab 90 mg | Group IV: Ustekinumab 45 mg Weekly for 4 Weeks | Group V: Ustekinumab 90 mg Weekly for 4 Weeks
Number analyzed (Participants) | 2 | 24 | 32 | 37 | 47
Particpants | 1 | 8 | 13 | 15 | 31

4. Secondary Outcome: Number of Participants Who Achieved Psoriasis Area Severity Index (PASI) 75% Improvement (0-72) at Week 28
Description: Psoriasis Area and Severity Index (PASI)(0 [ best] -72 [worst]) score at Week 28 for participants who were retreated at Week 16. This is a test of how bad a person's psoriasis is. The combination of redness, scaling, and thickness, as well as overall body involvement determine the PASI score.
Time Frame: Week 28
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Group I: Placebo | Group II: Ustekinumab 45 mg | Group III: Ustekinumab 90 mg | Group IV: Ustekinumab 45 mg Weekly for 4 Weeks | Group V: Ustekinumab 90 mg Weekly for 4 Weeks
Number analyzed (Participants) | 44 | 28 | 28 | 17 | 10
Participants | 29 | 8 | 18 | 8 | 3

ADVERSE EVENTS:
Time Frame: Week 36
Description: Three participants received placebo by mistake at Week 0, including 1 participant who was not randomized into the study and 2 participants who were randomized to a CNTO 1275 group but received the incorrect study agent. 1 participant not randomized but treated with placebo was included in the placebo group for adverse events
Groups:
- Placebo -> Ustekinumab 90 mg (After CP): After Controlled period (Week 20-36) - receiving placebo at Weeks 0, 1, 2, 3 and 16 -> receiving ustekinumab 90 mg at Week 20.
- Ustekinumab 45 mg (After CP): After Controlled period (Week 20-36) - receiving ustekinumab 45 mg at Week 0. At Week 16, participants with PGA >= 3 received ustekinumab 45 mg.
- Ustekinumab 90 mg (After CP): After Controlled period (Week 20-36) - receiving ustekinumab 90 mg at Week 0. At Week 16, participants with PGA >= 3 received ustekinumab 90 mg.
- Ustekinumab 45 mg Weekly for 4 Weeks (After CP): After Controlled period (Week 20-36) - receiving ustekinumab 45 mg at Weeks 0, 1, 2 and 3. At Week 16, participants with PGA >= 3 received ustekinumab 45 mg.
- Ustekinumab 90 mg Weekly for 4 Weeks (After CP): After Controlled period (Week 20-36) - receiving ustekinumab 90 mg at Weeks 0, 1, 2 and 3. At Week 16, participants with PGA >= 3 received ustekinumab 90 mg.
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP) | Ustekinumab 45 mg Weekly for 4 Weeks (CP) | Ustekinumab 90 mg Weekly for 4 Weeks (CP) | Placebo -> Ustekinumab 90 mg (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP) | Ustekinumab 45 mg Weekly for 4 Weeks (After CP) | Ustekinumab 90 mg Weekly for 4 Weeks (After CP)
Serious Adverse Events (participants affected / at risk) | 1/67 | 3/63 | 1/64 | 2/63 | 3/62 | 1/49 | 0/60 | 2/61 | 0/62 | 4/62
Other Adverse Events (participants affected / at risk) | 36/67 | 38/63 | 40/64 | 31/63 | 27/62 | 16/49 | 19/60 | 21/61 | 17/62 | 11/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=67) | Ustekinumab 45 mg (CP) (N=63) | Ustekinumab 90 mg (CP) (N=64) | Ustekinumab 45 mg Weekly for 4 Weeks (CP) (N=63) | Ustekinumab 90 mg Weekly for 4 Weeks (CP) (N=62) | Placebo -> Ustekinumab 90 mg (After CP) (N=49) | Ustekinumab 45 mg (After CP) (N=60) | Ustekinumab 90 mg (After CP) (N=61) | Ustekinumab 45 mg Weekly for 4 Weeks (After CP) (N=62) | Ustekinumab 90 mg Weekly for 4 Weeks (After CP) (N=62)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hernia congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzymes increased (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine fibroid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug dependence (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Psychosis (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Psoriasis aggravated (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral infarction (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=67) | Ustekinumab 45 mg (CP) (N=63) | Ustekinumab 90 mg (CP) (N=64) | Ustekinumab 45 mg Weekly for 4 Weeks (CP) (N=63) | Ustekinumab 90 mg Weekly for 4 Weeks (CP) (N=62) | Placebo -> Ustekinumab 90 mg (After CP) (N=49) | Ustekinumab 45 mg (After CP) (N=60) | Ustekinumab 90 mg (After CP) (N=61) | Ustekinumab 45 mg Weekly for 4 Weeks (After CP) (N=62) | Ustekinumab 90 mg Weekly for 4 Weeks (After CP) (N=62)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 4 | 1 | 0 | 1 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 4 | 1 | 3 | 1 | 2 | 1 | 2 | 5 | 3 | 1
Pain (Nervous system disorders) | 2 | 3 | 8 | 3 | 4 | 4 | 1 | 2 | 0 | 2
Headache (Nervous system disorders) | 11 | 12 | 12 | 2 | 9 | 0 | 2 | 3 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 4 | 4 | 2 | 1 | 1 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 4 | 1 | 4 | 1 | 1 | 0 | 2 | 0
Arthritis aggravated (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 4 | 3 | 1 | 0 | 2 | 1 | 1 | 0
Purpura (Blood and lymphatic system disorders) | 2 | 4 | 5 | 1 | 3 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 | 5 | 3 | 2 | 0 | 1 | 0 | 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 5 | 5 | 1 | 1 | 1 | 0 | 2 | 0
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 4 | 3 | 3 | 1 | 2 | 1 | 4 | 0
Upper resp tract infection (Respiratory, thoracic and mediastinal disorders) | 14 | 16 | 20 | 9 | 11 | 6 | 10 | 9 | 5 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 6 | 3 | 5 | 3 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The count of patients with any nonserious adverse events (NAE) excludes patients who only had NAE that occurred in <=5% of patients. This information may vary from existing approved labeling and publications due to the requirement of this website.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the only disclosure restriction on the PI is that the sponsor has 60 days to review results communications prior to public release and can embargo communications regarding trial results for a period that does not exceed 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.